CLINICAL TRIAL: NCT01532882
Title: Assessment of the Efficacy and Safety of Diosmin 600mg on Painful Symptomatology in Patients With Chronic Venous Disease of Lower Limbs: a Multicentric, Randomised, Double-blind, Placebo-controlled Trial in Parallel Groups
Brief Title: Efficacy and Safety of Diosmin 600mg Versus Placebo on Painful Symptomatology in Patients With Chronic Venous Disease of Lower Limbs
Acronym: EDEN
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Laboratoire Innotech International (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DIO401-10
Record Dates: First submitted 2012-02-10; First posted 2012-02-15 (Estimated); Last update posted 2013-04-29 (Estimated); Status verified 2013-04

CONDITIONS: Chronic Venous Disease of Lower Limbs
MeSH Terms: interventions — Diosmin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Diosmin (Experimental)
  Interventions: Drug: Diosmin
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Diosmin — tablet, 600mg, PO, 1 tab per day during 28 days
  Arms: Diosmin
Drug: Placebo — tablet, PO, 1 per day during 28 days
  Arms: Placebo

SUMMARY:
Diosmin has a well established use status in improvement of the symptoms of venolymphatic insufficiency: heavy legs, pain, primo-decubitus restlessness and as complement treatment of capillary fragility.

Nevertheless, diosmin 600 mg did not benefit from a rigorous clinical study versus placebo, to establish its efficacy in the pain relief in Chronic Venous Disease (CVD).

The aim of this project led by Dr. Guex is to evaluate the efficacy and safety of diosmin 600 mg - DIOVENOR® on the painful symptoms of CVD of the lower limbs, in a multicentre, controlled, randomised, double blind, placebo-controlled, parallel-group study.

ELIGIBILITY:
Inclusion Criteria:

1. Patient, man or woman, aged 18 and over,
2. Patient presenting a C1s or C2s venous disease grade of the lower limbs
3. Patient presenting a painful venous symptomatology in the lower limbs for at least 15 days.
4. Patient suffering from venous symptomatology in one leg with a painful symptom intensity higher or equal to 30 mm (VAS= 100mm)

Exclusion Criteria:

1. Patient treated by venotonic treatments or vascular protectants or assimilated dietary supplements or homeopathic treatments or diuretics within 15 days prior inclusion,
2. Patients who started treatments such as calcium inhibitors, beta-blockers, angiotensin converting enzyme inhibitors and/or vasodilators and/or vasoconstrictors within 28 days prior inclusion (for patients already taking this type of treatments, dosage should not have been changed in the 28 days prior inclusion and should not be planned to change in the course of the study),
3. Patient treated by any analgesic within 7 days prior inclusion,
4. Patient treated by an anti-inflammatory treatment within 7 days prior inclusion,
5. Patient using elastic venous compression
6. Patient presenting permanent oedema,
7. Patients presenting venous skin changes,
8. Patient whose activity in the 4 following weeks (that is to say during the study) would be different from his/her usual activities (before the study),
9. Patient suffering from a pathology generating other pains than venous pains in the lower limbs,
10. Patient with a history of lower limbs trauma responsible for sequel pains,
11. Patient with a known deep venous reflux,
12. Patient with a history of venous thromboses or thrombo-embolic diseases within the last 6 months before inclusion,
13. Patient treated with analgesics or anti-inflammatory treatments used as analgesics within 4 weeks prior inclusion
14. Patient having a known hypersensitivity to diosmin or one of the excipients
15. Patients with rare hereditary problems of galactose intolerance, the Lapp lactase deficiency or glucose-galactose malabsorption ),

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 378 (Actual)
Dates: Start 2012-01; Primary Completion 2013-03 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Change of Visual analog Scale score for assessment of the painful venous symptomatology | baseline and after 28 days

SECONDARY OUTCOMES:
- Painful symptom intensity (daily VAS score) Area Under the Curve | 28 days
- Daily VAS score for Response rate | 28 days
- Daily VAS score for Time to response | 28 days
- Score of Quality of life questionnaire (SQOR-V) | Between baseline and 28 days
- Patient's and physician's global satisfaction score | At 28 days
Adverse Events (numbers and frequency) | 28 days
- Unusual intakes of analgesic treatments (rate of patients) | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Jérôme GUEX, MD, Principal Investigator
Locations (1):
- Dr Jean-Jérôme GUEX, Nice, France

REFERENCES:
- [Derived] Martinez-Zapata MJ, Vernooij RW, Simancas-Racines D, Uriona Tuma SM, Stein AT, Moreno Carriles RMM, Vargas E, Bonfill Cosp X. Phlebotonics for venous insufficiency. Cochrane Database Syst Rev. 2020 Nov 3;11(11):CD003229. doi: 10.1002/14651858.CD003229.pub4. PMID 33141449